CLINICAL TRIAL: NCT05008458
Title: Value of Von Willebrand Factor and Copeptin Assay in Children With Febrile Seizures at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Ali Abdelrady, resident doctor at pediateric department sohag university hospital, Sohag University
Other Study IDs: soh-med-21-07-16
Record Dates: First submitted 2021-07-28; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Febrile Seizure
MeSH Terms: conditions — Seizures, Febrile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- children with febrile seizures
  Interventions: Diagnostic Test: von willebrand factor and copeptin
- febrile children without seizures
  Interventions: Diagnostic Test: von willebrand factor and copeptin
- healthy control children
  Interventions: Diagnostic Test: von willebrand factor and copeptin

INTERVENTIONS:
Diagnostic Test: von willebrand factor and copeptin — biomarkers increase in children with febrile seizures

SUMMARY:
Febrile seizures are one of the most common clinical diseases in pediatric neurology. It occurs between 6 months and 6 years of age and occurs in ~2-5% of children. According to the age, frequency, duration, and type of seizures FS is divided into simple febrile seizures and complex febrile seizures Differentiation between febrile seizures and non-ictal events associated with fever such as shivering or dizziness is challenging. Therefore, precise diagnosis of FS after paroxysmal episodes associated with fever is often hindered by the lack of an objective biomarker With the widespread application of technologies, such as molecular biology, in medicine, some biomarkers for predicting or diagnosing FS have attracted attention. Imuekemhe et al in 1989 and 1996 found that lactic acid in the serum and cerebrospinal fluid of children with FS was significantly increased . Arginin-vasopressin hormone AVP released by the pituitary gland, has been shown to be involved in the thermoregulatory response to fever and convulsions Although AVP is unstable in the peripheral blood and, therefore, unsuited for diagnostic use the C-terminal portion of the AVP precursor copeptin has been recognized as a robust marker of AVP secretion . Wellman et al. found that the serum copeptin and Von Willebrand factor of children with FS were significantly higher than those of the control group .

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 months to 6 years.
* Seizures.
* Fever (≥38°C).

Exclusion Criteria:

* Central nervous system infection.
* Epilepsy.
* Previous neurological abnormalities.
* Inborn errors of metabolism.
* Immunological diseases.
* Endocrinal diseases (e.g., diabetes mellitus).
* Obesity.
* Eating disorders.
* Gastrointestinal disorders (e.g., diarrhea).

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include three groups of children (30 for each): children with febrile seizures (group 1), febrile children without seizures (group 2), and healthy control children (group 3).
  at Pediatric neurology outpatient clinic and Pediatric Department at Sohag University Hospital.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Value of von willebrand factor and copeptin assay in children with febrile seizures at Sohag University Hospital | one year
  Serum copeptin and Von Willebrand factor (VWF) venous blood samples (3 ml) will be obtained from children with FS (within 3 hours of seizures) as well as the two control groups. .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Patel N, Ram D, Swiderska N, Mewasingh LD, Newton RW, Offringa M. Febrile seizures. BMJ. 2015 Aug 18;351:h4240. doi: 10.1136/bmj.h4240. No abstract available. PMID 26286537
- [Background] Leung AK, Hon KL, Leung TN. Febrile seizures: an overview. Drugs Context. 2018 Jul 16;7:212536. doi: 10.7573/dic.212536. eCollection 2018. PMID 30038660
- [Background] Pechmann A, Wellmann S, Stoecklin B, Kruger M, Zieger B. Increased von Willebrand factor parameters in children with febrile seizures. PLoS One. 2019 Jan 3;14(1):e0210004. doi: 10.1371/journal.pone.0210004. eCollection 2019. PMID 30605489